CLINICAL TRIAL: NCT01827176
Title: Clinical Characteristic of Recurrent Acute Rhinosinusitis in Children
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, JITTIMA VESKITKUL, Dr., Mahidol University
Other Study IDs: 094/2556(EC4)
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Recurrent Sinusitis
Keywords: Characteristic; Recurrent Acute Rhinosinusitis; Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Recurrent Acute Rhinosinusitis: Recurrent Acute Rhinosinusitis is defined as acute rhinosinusitis more than 3 times/6 months or more than 4 times/year
  Interventions: Other: Recurrent Acute Rhinosinusitis

INTERVENTIONS:
Other: Recurrent Acute Rhinosinusitis — Clinical Characteristic of Recurrent Acute Rhinosinusitis

SUMMARY:
The purpose of this study is to determine the clinical characteristic of recurrent acute rhinosinusitis in children.

ELIGIBILITY:
Inclusion Criteria:

* Children the age less than 15 years with recurrent acute rhinosinusitis who are attending the pediatric allergy clinic during Jan 2010 - Dec 2012.

Exclusion Criteria:

* Children who had lost medical record.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients from pediatric allergy clinic will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Presenting symptoms of recurrent acute rhinosinusitis | 12 months

SECONDARY OUTCOMES:
Age of onset | 12 months

OTHER OUTCOMES:
Number of sinusitis after received treatment | 12 months
Immunological profile | 12 months
  immunoglobulin level and immunoglobulin G subclass level
Number of participants with allergic rhinitis | 12 months
Number of participants with immunodeficiency | 12 months
Number of participants with adenotonsillar hypertrophy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jittima Veskitkul, MD, Principal Investigator — Mahidol University
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Veskitkul J, Vichyanond P, Pacharn P, Visitsunthorn N, Jirapongsananuruk O. Clinical characteristics of recurrent acute rhinosinusitis in children. Asian Pac J Allergy Immunol. 2015 Dec;33(4):276-80. doi: 10.12932/AP0591.33.4.2015. PMID 26708390